CLINICAL TRIAL: NCT05797571
Title: Informal Caregivers and Clinicians' Knowledge, Awareness, Attitude and Expect Barriers Towards Internet-based Interventions: A Stakeholders' Survey in Italy
Brief Title: SOSteniamoci: Stakeholders' Survey
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 03C212
Record Dates: First submitted 2023-03-13; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Informal Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Informal care is defined as the unpaid care provided to an older, frail, or ill person, by a person such as a spouse, a parent, a child, another relative, a neighbor, or a friend. This phenomenon may lead to stress, burden, and decreased informal caregivers' quality of life. Since lack of time, distance from services, and financial strains make the provision of psychological interventions to informal caregivers often challenging, Internet-based (self-help) programs might represent a viable solution to promote their emotional well-being. Still, despite the proven benefits of internet-based intervention, no available programs for informal caregivers are available for the Italian population. Nevertheless, planning and developing an online intervention, involving possible stakeholders (caregivers), might facilitate the understanding and dissemination of, willingness to use, and success of the future intervention. Thus, the goal of the current study is to assess Italian stakeholders' knowledge about, awareness of, attitudes towards, willingness to participate and use, and expected barriers to internet-based interventions.

DETAILED DESCRIPTION:
The present study assessed the knowledge and awareness, attitudes, willingness to participate in, and expected barriers towards using Internet-based interventions to alleviate caregivers' burden in a sample of Italian caregivers and clinicians. To this aim, an online stakeholders' survey was conducted in Italy among clinicians and informal caregivers, using a snowballing sampling technique. Participants were asked to fill in the informed consent and complete the online survey as a clinician, a caregiver, or both. Data were monitored daily. Descriptive statistics and Pearson correlation analysis were used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinicians and informal caregivers
* aged 18 years or older
* internet access
* basic computer literacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Formal and informal caregivers
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Mean score in Online survey for clinicians | At baseline, during online survey, performed after signing informed consent
  Online survey for clinicians - 30 items
Mean score in Online survey for informal caregivers | At baseline, during online survey, performed after signing informed consent
  Online survey for informal caregivers - 45 items

CONTACTS AND LOCATIONS:
Overall Officials: Giada Pietrabissa, PhD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Giada Pietrabissa, Milan, Italy